CLINICAL TRIAL: NCT05124080
Title: An Investigator Initiated Open Label Study Evaluating the Efficacy and Tolerability of Oral Deucravacitinib for the Treatment of Nail Psoriasis
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Boni Elewski, Professor, University of Alabama at Birmingham
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-300008245; 2028180 (Other Grant/Funding Number: Bristol Myers Squibb)
Record Dates: First submitted 2021-11-05; First posted 2021-11-17 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2025-12

CONDITIONS: Nail Psoriasis
MeSH Terms: interventions — deucravacitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Deucravacitinib 6 mg Daily (Experimental): All participants will receive 6 mg of deucravacitinib daily.
  Interventions: Drug: Deucravacitinib

INTERVENTIONS:
Drug: Deucravacitinib — All participants will receive 6 mg of Deucravacitinib daily.

SUMMARY:
. An open label proof of concept study will be conducted to assess the efficacy and safety of deucravactinib for treatment of nail psoriasis. Twenty adult patients with nail psorasis and skin disease qualifying for a systemic agent per investigator will be treated with deucravacitinib 6 mg daily. Subjects will be assessed for a total of 48 weeks. Psoriasis assessments such as the modified Nail Psoriasis Severity Index will be conducted. Photos will be used to document nail involvement. Descriptive statistical analysis will be conducted at the conclusion of the study.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 and older
* Give written informed consent prior to any study procedures being conducted, and candidates will authorize the release and use of protected health information (PHI)
* Be willing and consent to having photos taken of their fingernails
* Must be in general good health (except for disease under study) as judged by the Investigator, based on medical history, physical examination, clinical laboratories, and urinalysis. (NOTE: The definition of good health means a subject does not have uncontrolled significant co-morbid conditions).
* Diagnosis of chronic plaque psoriasis that has been present for at least 6 months prior to baseline
* Plaque psoriasis qualifying for a systemic agent per investigator.
* Nail psoriasis in at least one finger nail with a mNAPSI of 8 or greater or a total modified Nail Psoriasis Severity Index of 20 or greater
* A Nail Pain NRS score of 3 or higher. The Nail Pain NRS will assess the severity of pain linked to the nail disease.
* Must have discontinued all systemic therapies for the treatment of psoriasis or psoriatic arthritis at least 4 weeks or 5 half-lives, and biologics for at least 2 months or 5 half-lives (whichever is longer) prior to baseline visit
* Must have discontinued all topical therapies for the treatment of psoriasis at least 2 weeks prior to baseline visit
* Subjects must have discontinued UV therapy at least 2 weeks prior to baseline and PUVA at least 4 weeks prior to baseline.
* Subjects must be in good general health without significant uncontrolled comorbidities, other than psoriasis, as determined by the investigator based on exam findings, medical history, and clinical laboratories. Patients with stable mild renal insufficiency are eligible for enrolling in this trial.
* Females of childbearing potential must use an approved birth control method while receiving treatment and for 28 days following the last dose of deucravacitinib, and there must be a documented negative pregnancy tests prior to initiating treatment. Approved birth control methods include hormonal contraception (oral, injection, implant, transdermal patch, vaginal ring), intrauterine device, tubal ligation (tying your tubes), partners vasectomy, or male or female condoms that are not made of natural materials PLUS a diaphragm with spermicide, cervical cap with spermicide, or a contraceptive sponge with spermicide. Females not of child bearing potential are defined as being at least 1 year postmenopausal or surgically sterile (bilateral tubal ligation, bilateral oophorectomy and/or hysterectomy).
* Male subjects, including those who have had a vasectomy, must use condoms not made of natural materials for the duration of the trial and for at least 28 days after the last dose of deucravacitinib if conception is possible.

Exclusion Criteria:

* Other than disease under study, any clinically significant (as determined by the Investigator) cardiac, endocrinologic, pulmonary, neurologic, psychiatric, hepatic, renal, hematologic, immunologic disease, or other major disease that is currently uncontrolled.
* Any condition, including the presence of laboratory abnormalities, which would place the subject at unacceptable risk if he/she were to participate in the study.
* Prior history of suicide attempt at any time in the subject's life time prior to screening or randomization, or major psychiatric illness requiring hospitalization within the last 3 years.
* Pregnant or breast feeding.
* Active substance abuse or a history of substance abuse within 6 months prior to Screening.
* Malignancy or history of malignancy, except for:

  1. treated [ie, cured] basal cell or squamous cell in situ skin carcinomas;
  2. treated [ie, cured] cervical intraepithelial neoplasia (CIN) or carcinoma in situ of cervix with no evidence of recurrence within the previous 5 years.
* Use of any investigational drug within 4 weeks prior to randomization, or 5 pharmacokinetic/pharmacodynamic half lives, if known (whichever is longer).
* Prior treatment with deucravacitinib.
* Unable to comply with the protocol (as defined by the Investigator; i.e. drug or alcohol abuse or history of noncompliance).
* Concomitant therapy with medications that are strong cytochrome P450 inducers, including rifampin, phenobarbital, carbamazepine, or phenytoin.
* Any other dermatologic conditions that prohibit or confound the ability of the investigator to interpret skin and/or nail exam findings.
* Patients who will be unable to avoid the use of systemic steroids, excluding intranasal or inhaled steroids that will be permitted, for the duration of the trial.
* Any known hypersensitivity to deucravacitinib.
* Prisoners or subjects who are involuntarily incarcerated
* Subjects who are compulsorily detained for treatment of either psychiatric or physical illness
* Inability to comply with restrictions and prohibited activities listed in study protocol
* Site personnel or their immediate family

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2024-03-01 (Actual); Primary Completion 2025-12-01 (Actual); Study Completion 2025-12-01 (Actual)

PRIMARY OUTCOMES:
Change in the modified Nail Psoriasis Severity Index (mNAPSI) compared to baseline | baseline to week 24
  Mean percent change of mNAPSI

CONTACTS AND LOCATIONS:
Locations (1):
- University of Alabama at Birmingham - Department of Dermatology, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No